CLINICAL TRIAL: NCT03090464
Title: A Real-world, Point-of-care, Randomized, Parallel Group, Open, 6-month Clinical Study to Evaluate the Effect of a Digital Disease Management Tool in Patients With Type 2 Diabetes Mellitus
Brief Title: A 6-month Clinical Study to Evaluate the Effect of a Digital Disease Management Tool in Patients With T2DM
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1841C00004
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Digital disease management; T2DM; Hyperglycemia; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard of Care (SOC): Participants have standard of care with no access to digital disease management tool
- SOC + digital disease management: Participants have access to the digital disease management tool in addition to standard of care
  Interventions: Other: Use of digital disease management tool

INTERVENTIONS:
Other: Use of digital disease management tool — The purpose of the study is to evaluate if the provision of a digital disease management tool, in addition to SOC for T2DM, will improve glycemic control. The impact of the tool will be assessed in comparison to a Control group who will receive SOC alone. All participants will complete the PRO assessments. This is a real world study carried out at the point of care.
  Groups: SOC + digital disease management

SUMMARY:
Type 2 diabetes mellitus is a complex, chronic disease that requires a comprehensive treatment plan aimed at meeting multitude therapeutic targets associated with micro- and macro-vascular risk reduction. There is evidence that patient support in various forms can have a significant positive impact on adherence to treatment and the meeting of targets in patients with type 2 diabetes mellitus. The purpose of this study is to evaluate if the use of a digital disease management tool (Smart phone- web portal-based tool), in addition to Standard of Care for T2DM, will improve glycemic control. Other variables important in T2DM (such as weight, blood pressure, and lipid levels), will also be evaluated along with patient-reported outcomes, such as satisfaction with treatment and adherence to their antihyperglycemic treatment. Study duration is 6 months

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a complex, chronic disease that requires a comprehensive treatment plan aimed at meeting multitude therapeutic targets associated with micro- and macro-vascular risk reduction. There is evidence that patient support in various forms can have a significant positive impact on adherence to treatment and the meeting of targets in patients with type 2 diabetes mellitus. A digital disease-management tool, smart phone- and web-based portal, has been developed that incorporates the following features aimed at improving patient and population outcomes:

Treatment management to help patients remember to take medications and track adherence; Goal setting, including medical nutrition therapy, appropriately prescribed physical activity, and weight loss for those patients who are overweight or obese; Tracking and data collection for blood glucose, weight, and exercise, as entered by the patient or automatically for activity via Bluetooth pedometer or activity tracker; Assessments to capture patient beliefs in order to tailor personalized content to individual needs; educational and motivational content in the form of short messages, text, and videos covering T2DM and its treatment, and lifestyle advice; Web portals to display collected data back to the patient and healthcare practitioner in real-time to allow better and timely management of diabetes.

This tool is added to the Standard of Care for T2DM. Data are collected for patients utilizing this tool, compared with those who are not. Clinical assessments as part of the Standard of Care are collected, as well as standard Patient Reported Outcomes for this disease.

Glycemic control is considered to be the goal of a T2DM disease management plan.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent;
* Diagnosed with T2DM;
* Male or female aged >/= 18 years at time of consent;
* Treatment with 1 or more non-insulin antihyperglycemic medications for at least 6 months prior to enrollment;
* Own or have access to a smart phone with internet access and have access to the internet via a tablet or personal computer at least once a day;
* HbA1c levels must be obtained at the enrollment visit or up to 14 days prior to Visit 1 and must be >/=7.5% and </=11.0%. Most of the hbA1c values obtained within the past 9 months must also be within this range;
* Body mass index >/= 25 and </=55 kg/mm2 within the last 3 months;
* Ability to communicate in English;
* Judged by their primary care physician to have suitable hearing, vision, manual dexterity, ability to understand instructions, and ability to use and understand smart phone and internet applications;
* Negative pregnancy test for female subjects of childbearing potential.

Exclusion Criteria:

* Pregnancy;
* Insulin use at baseline;
* Current use of a smart phone- or web portal-based tool designed to help with management of T2DM;
* History of Type 1 diabetes or ketoacidosis;
* Currently taking weight loss medication;
* Involvement in the planning and/or conduct of this study;
* Previous enrollment in the present study;
* Participation in a clinical study with an investigational product or a disease state management program during the last 30 days;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 diabetes mellitus who are on 1 or more non-insulin antihyperglycemic medications for at least 6 months prior to enrollment.
Sampling Method: Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of study (Month 6) in HbA1c levels | 6 months
  Assessed from blood samples taken at visits per standard of care

SECONDARY OUTCOMES:
Percentage of patients who achieve HbA1c levels <7% at Month 6 | 6 Months
  Assessed from blood samples taken at visits per standard of care
Mean change in body weight (kg) from baseline to Month 6 | 6 Months
  Measures taken at visits per standard of care
Proportion of patients in both cohorts who intensify antihyperglycemic treatment from Visit 1 | 6 Months
  Defined as an increase in dose or addition of a new antihyperglycemic agent not received at baseline

OTHER OUTCOMES:
Number of times the smart phone- and/or web portal-based tool is accessed per patient | 6 Months
  Calculated by adding the total number of discrete log-in attempts to the tool for each patient using the tool at least once
Length of time from first to last usage of smart phone- and/or web portal-based tool across the course of the study | 6 Months
  Determined by calculating the time from first to last log-in attempt for each patient accessing the tool at least twice during the course of the study
Mean patient satisfaction with the digital disease management tool | 6 Months
  Assessed by the User Satisfaction Survey
Mean percent change from baseline to Month 6 in systolic blood pressure | 6 Months
  Measures taken at visits per standard of care
Mean percent change from baseline to Month 6 in low-density lipoprotein-cholesterol (LDL-C) | 6 Months
  Assessed from blood samples taken at visits per standard of care
Percent of patients who achieve blood pressure <140/90 mmHg at Month 6 | 6 Months
  Measures taken at visits per standard of care
Percent of patients who achieve LDL-C <100 mg/dL at Month 6 | 6 Months
  Assessed from blood samples taken at visits per standard of care
Differences in primary care office visits between active and control group during the 6-month study period | 6 Months
  As reported in patient records
Differences in Emergency Room visits between active and control group during the 6-month study period as reported in patients at the end of the study | 6 Months
  As reported by patients at the end of the study
Change in baseline to Month 6 in Diabetes Treatment Satisfaction Questionnaire - Status version score | 6 Months
  As assessed in the Patient Reported Outcome measure Diabetes Treatment Satisfaction Questionnaire - Status version at the point-of-care visits
Change in baseline to Month 6 in Diabetes Self-Management Questionnaire score (16-question) (patient perception on ability to manage their disease) | 6 Months
  As assessed in the Patient Reported Outcomes measure Diabetes Self-Management Questionnaire at the point-of-care visits
Change in baseline to Month 6 in Morisky Medication Adherence Scale (8-item) (adherence) | 6 Months
  As assessed in the Patient Reported Outcome measure Morisky Medication Adherence Scale at the point-of-care visits

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Sooben, Study Chair — AstraZeneca
Locations (44):
- United States (44):
  - Research Site, Birmingham, Alabama
  - Research Site, Peoria, Arizona
  - Research Site, Surprise, Arizona
  - Research Site, Lincoln, California
  - Resezrch Site, Montclair, California
  - Research Site, North Hollywood, California
  - Research Site, Spring Valley, California
  - Research Site, Van Nuys, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Cooper City, Florida
  - Research Site, DeLand, Florida
  - Research Site, Hialeah, Florida
  - Reserarch Site, Jacksonville, Florida
  - Research Site, Lake City, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Tampa, Florida
  - Research Site, Evanston, Illinois
  - Research Site, Lexington, Kentucky
  - Research Site, Oxon Hill, Maryland
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, New Windsor, New York
  - Research Site, Westfield, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Franklin, Ohio
  - Research Site, Downingtown, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Tullahoma, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Lampasas, Texas
  - Research Site, Plano, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Burke, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Federal Way, Washington
  - Research Site, Olympia, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14670&filename=D1841C00004%20CSR%20synopsis%20v1.0%2022OCT2018%20redacted.pdf